CLINICAL TRIAL: NCT02471404
Title: A 52-Week, Multi-Centre, Randomised, Parallel-Group, Double-Blind, Active Controlled, Phase IV Study to Evaluate the Safety and Efficacy of Dapagliflozin or Dapagliflozin Plus Saxagliptin Compared With Sulphonylurea All Given as Add-on Therapy to Metformin in Adult Patients With Type 2 Diabetes Who Have Inadequate Glycaemic Control on Metformin Monotherapy
Brief Title: Efficacy and Safety of Dapagliflozin and Dapagliflozin Plus Saxagliptin in Combination With Metformin in Type 2 Diabetes Patients Compared With Sulphonylurea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D1689C00014
Record Dates: First submitted 2015-06-11; First posted 2015-06-15 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus; Inadequate Glycaemic Control
Keywords: Diabetes Mellitus Type 2,; metformin,; saxagliptin,; dapagliflozin,; glimepiride,; inadequate glycaemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; saxagliptin; glimepiride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dapagliflozin+metformin (Active Comparator): Dapagliflozin + saxagliptin placebo + glimepiride placebo + metformin
  Interventions: Drug: Dapagliflozin; Drug: Placebo for saxagliptin; Drug: Placebo for glimepiride
- Dapagliflozin+saxagliptin+metformin (Active Comparator): Dapagliflozin + saxagliptin + glimepiride placebo+ metformin
  Interventions: Drug: Dapagliflozin; Drug: Saxagliptin; Drug: Placebo for glimepiride
- Glimepiride+metformin (Active Comparator): Glimepiride + dapagliflozin placebo + saxagliptin placebo + metformin
  Interventions: Drug: Glimepiride; Drug: Placebo for dapagliflozin; Drug: Placebo for saxagliptin

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg, orally Green, plain, diamond-shaped, film-coated tablet
  Other Names: Forxiga
  Arms: Dapagliflozin+metformin; Dapagliflozin+saxagliptin+metformin
Drug: Saxagliptin — 5 mg, orally Plain, yellow, biconvex, round, film-coated tablet
  Other Names: Onglyza™
  Arms: Dapagliflozin+saxagliptin+metformin
Drug: Glimepiride — 1, 2, or 4 mg, orally Opaque gray capsule
  Other Names: Amaryl
  Arms: Glimepiride+metformin
Drug: Placebo for dapagliflozin — Does not contain active ingredient, orally Green, plain, diamond-shaped, film-coated tablet
  Arms: Glimepiride+metformin
Drug: Placebo for saxagliptin — Does not contain active ingredient, orally Plain, yellow, biconvex, round, film-coated tablet
  Arms: Dapagliflozin+metformin; Glimepiride+metformin
Drug: Placebo for glimepiride — Does not contain active ingredient, orally. Opaque gray capsule
  Arms: Dapagliflozin+metformin; Dapagliflozin+saxagliptin+metformin

SUMMARY:
This study is being carried out to see if dapagliflozin and dapagliflozin plus saxagliptin as an addition to metformin is effective and safe in treating patients with type 2 diabetes when compared to glimepiride (sulphonylurea) as an addition to metformin treatment.

ELIGIBILITY:
Inclusion Criteria: Main Inclusion Criteria:

1. Is male or female and ≥18 and <75 years old at time of informed consent.
2. Has a HbA1c of ≥7.5% and ≤10.5% based on central laboratory results from Visit 1, with individual need for therapy escalation.
3. Currently treated with a stable maximum tolarated dose (MTD) (≥1500 mg/day) of metformin therapy for at least 8 weeks prior to Enrolment visit.
4. Has a BMI of ≤45 kg/m2 at Enrolment visit.
5. Has a C-peptide laboratory value of ≥1.0 ng/mL (0.33 nmol/L; 333.3 pmol/L) based on central laboratory results from Visit 1.

Main, Exclusion Criteria:

1. Clinically diagnosed with Type I diabetes, known diagnosis of maturity onset diabetes of the young (MODY), or secondary diabetes mellitus or known presence of glutamate decarboxylase 65 (GAD65) antibodies.
2. Patients who, in the judgment of the Investigator, may be at risk for dehydration or volume depletion that may affect the patient's safety and/or the interpretation of efficacy or safety data.
3. Clinically significant cardiovascular disease or procedure within 3 months prior to Enrolment or expected to require coronary revascularization procedure during the course of the study.
4. Concomitant treatment with loop diuretics

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 939 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2017-03-13 (Actual); Study Completion 2017-03-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (145):
- Czechia (10):
  - Research Site, Hodonín
  - Research Site, Hradec Králové
  - Research Site, Jílové u Prahy
  - Research Site, Ostrava - Belsky Les
  - Research Site, Pardubice
  - Research Site, Plzen - Severni Predmesti
  - Research Site, Praha Klanovice
  - Research Site, Přelouč
  - Research Site, Uherské Hradiště
  - Research Site, Zlín
- Germany (90):
  - Research Site, Aschaffenburg
  - Research Site, Bad Homburg
  - Research Site, Bad Mergentheim
  - Research Site, Bad Nauheim
  - Research Site, Bad Neuenahr-Ahrweiler
  - Research Site, Bad Oeynhausen
  - Research Site, Bad Reichenhall
  - Research Site, Berlin
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Bünde
  - Research Site, Cologne
  - Research Site, Daaden
  - Research Site, Darmstadt
  - Research Site, Datteln
  - Research Site, Deggingen
  - Research Site, Dippoldiswalde
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Eschweiler
  - Research Site, Essen
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Freudenstadt
  - Research Site, Gelnhausen
  - Research Site, Giengen an der Brenz
  - Research Site, Goch
  - Research Site, Göttingen
  - Research Site, Grevesmühlen
  - Research Site, Großheirath
  - Research Site, Hamburg
  - Research Site, Hamelin
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, Hildesheim
  - Research Site, Hof
  - Research Site, Hohenmölsen
  - Research Site, Höhenkirchen
  - Research Site, Jerichow
  - Research Site, Kallstadt
  - Research Site, Karlsruhe
  - Research Site, Kassel
  - Research Site, Kiel-Kronshagen
  - Research Site, Köthen
  - Research Site, Leipzig
  - Research Site, Lichtenfels
  - Research Site, Lingen
  - Research Site, Löhne
  - Research Site, Ludwigshafen
  - Research Site, Magdeburg
  - Research Site, Mannheim
  - Research Site, Marburg
  - Research Site, Marl
  - Research Site, Meine
  - Research Site, Meißen
  - Research Site, Mühldorf A. Inn
  - Research Site, München
  - Research Site, Münster
  - Research Site, Neumünster
  - Research Site, Neuwied Am Rhein
  - Research Site, Oldenburg
  - Research Site, Papenburg
  - Research Site, Pirna
  - Research Site, Rehburg-Loccum
  - Research Site, Rehlingen-Siersburg
  - Research Site, Reinfeld
  - Research Site, Remagen
  - Research Site, Rhaunen
  - Research Site, Rodgau-Dudenhofen
  - Research Site, Saarlouis
  - Research Site, Schwabenheim
  - Research Site, Speyer
  - Research Site, Stadtbergen
  - Research Site, Stolberg
  - Research Site, Straubing
  - Research Site, Stuttgart
  - Research Site, Sulzbach
  - Research Site, Trier
  - Research Site, Villingen-Schwenningen
  - Research Site, Wahlstedt
  - Research Site, Wangen
  - Research Site, Weinheim
  - Research Site, Westerkappeln
  - Research Site, Wetzlar
  - Research Site, Witten
- Hungary (15):
  - Research Site, Ács
  - Research Site, Budapest
  - Research Site, Csongrád
  - Research Site, Debrecen
  - Research Site, Esztergom
  - Research Site, Hatvan
  - Research Site, Kisvárda
  - Research Site, Komárom
  - Research Site, Miskolc
  - Research Site, Mosonmagyaróvár
  - Research Site, Nyíregyháza
  - Research Site, Orosháza-Szentetornya
  - Research Site, Pécs
  - Research Site, Polgár
  - Research Site, Székesfehérvár
- Poland (14):
  - Research Site, Bochnia
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Gdansk
  - Research Site, Koluszki
  - Research Site, Krakow
  - Research Site, Legnica
  - Research Site, Lodz
  - Research Site, Mrągowo
  - Research Site, Ostrowiec Świętokrzyski
  - Research Site, Poznan
  - Research Site, Sobótka
  - Research Site, Wierzchosławice
  - Research Site, Wroclaw
- Slovakia (16):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Lučenec
  - Research Site, Malacky
  - Research Site, Námestovo
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Prievidza
  - Research Site, Púchov
  - Research Site, Rimavská Sobota
  - Research Site, Sabinov
  - Research Site, Trenčín
  - Research Site, Trnava
  - Research Site, Vrútky

REFERENCES:
- [Derived] Muller-Wieland D, Kellerer M, Cypryk K, Skripova D, Rohwedder K, Johnsson E, Garcia-Sanchez R, Kurlyandskaya R, Sjostrom CD, Jacob S, Seufert J, Dronamraju N, Csomos K. Efficacy and safety of dapagliflozin or dapagliflozin plus saxagliptin versus glimepiride as add-on to metformin in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Nov;20(11):2598-2607. doi: 10.1111/dom.13437. Epub 2018 Jul 16. PMID 29947099
- See also: d1689c00014_SAP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3910&filename=d1689c00014_SAP_Redacted.pdf
- See also: d1689c00014_CSP_Redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3910&filename=d1689c00014_CSP_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Dapagliflozin 10mg: Dapagliflozin 10mg + Metformin
- Saxagliptin 5mg and Dapagliflozin 10mg: Saxagliptin 5mg and Dapagliflozin 10mg + Metformin
- Glimepiride 1mg/2mg/4mg: Glimepiride 1mg/2mg/4mg + Metformin
Period: Overall Study
Arm/Group | Dapagliflozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Started | 314 | 312 | 313
Completed | 281 | 298 | 288
Not Completed | 33 | 14 | 25
Not completed — Adverse Event | 7 | 1 | 2
Not completed — Developed Study Withdrawal Criteria | 4 | 1 | 2
Not completed — Failure to Meet Randomization Criteria | 2 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 3
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 4 | 5
Not completed — Other reasons not specified | 10 | 7 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg | Total
Number analyzed (Participants) | 314 | 312 | 313 | 939
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.4 (9.36) [31 to 75] | 59.2 (7.87) [36 to 74] | 58.6 (8.38) [34 to 75] | 58.4 (8.58) [31 to 75]
Age, Customized [Number; unit: Participants]
  <65 | 232 | 226 | 226 | 684
  >=65-<75 | 81 | 86 | 85 | 252
  >=75 | 1 | 0 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 122 | 105 | 339
  Male | 202 | 190 | 208 | 600
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 3 | 0 | 4
  Black Or African American | 2 | 2 | 2 | 6
  White | 311 | 307 | 311 | 929

OUTCOME MEASURES:

1. Primary Outcome: Change in Haemoglobin A1c (HbA1c) From Baseline to Week 52
Description: Change in HbA1c from baseline (week 0) to week 52.
Time Frame: Baseline, week 52. Values recorded after rescue treatment or collected more than 8 days after the last dose date were excluded from the analysis
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: HbA1c %
Groups:
- Dapaglifozin 10mg: Dapaglifozin 10mg + Metformin
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
HbA1c % | -0.82 (0.049) | -1.2 (0.046) | -0.99 (0.048)
Statistical Analysis 1: Comparison: Dapaglifozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Non-Inferiority — The non-inferiority (NI) margin was determined to be 0.30% (in absolute terms). A difference of ≤0.30%, in HbA1c change from b/l to wk 52 between the treatment groups was considered clinically equivalent. NI was assessed using the 2-sided 95% CI of adjusted mean difference between dapagliflozin or dapagliflozin plus saxagliptin and glimepiride; Mixed Models Analysis; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.0294 to 0.2986]
Statistical Analysis 2: Comparison: Saxagliptin 5mg and Dapagliflozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Non-Inferiority — The non-inferiority (NI) margin was determined to be 0.30% (in absolute terms). A difference of ≤0.30%, in HbA1c change from b/l to wk 52 between the treatment groups was considered clinically equivalent. NI was assessed using the 2-sided 95% Confidence Interval of adjusted mean difference between dapagliflozin or dapagliflozin plus saxagliptin and glimepiride; p = 0.001, Mixed Models Analysis — (superiority); Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.3443 to -0.0825]

2. Secondary Outcome: Patients With at Least One Episode of Confirmed Hypoglycaemia
Description: Percentage of patients reporting at least 1 episode of hypoglycaemia (symptomatic + blood glucose <=50 mg/dL) during the double-blind treatment period
Time Frame: Up to Week 52. Values recorded after rescue treatment or collected more than 8 days after the last dose date were excluded from the analysis
Population: Full Analysis Set
Measure: Number; unit: Percentage of participants
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
Percentage of participants | 0 | 0.32 | 4.21
Statistical Analysis 1: Comparison: Dapaglifozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Fisher Exact; Risk Difference (RD) = -4.21, 95% CI 2-sided [-6.45 to -1.97], Standard Error of Mean 1.14
Statistical Analysis 2: Comparison: Saxagliptin 5mg and Dapagliflozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Fisher Exact; Risk Difference (RD) = -3.89, 95% CI 2-sided [-6.21 to -1.56], Standard Error of Mean 1.19

3. Secondary Outcome: Change in Total Body Weight From Baseline at Week 52
Description: Change in body weight from baseline (week 0) to week 52
Time Frame: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Weight (kg)
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
Weight (kg) | -3.54 (0.231) | -3.15 (0.219) | 1.76 (0.224)
Statistical Analysis 1: Comparison: Dapaglifozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -5.30, 95% CI 2-sided [-5.93 to -4.67]
Statistical Analysis 2: Comparison: Saxagliptin 5mg and Dapagliflozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -4.91, 95% CI 2-sided [-5.52 to -4.29]

4. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 52
Description: Change in FPG from baseline (week 0) to week 52
Time Frame: as for outcome 1
Population: Full Analysis Set
Measure: Least Squares Mean (Standard Error); unit: FPG (mmol/L)
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
FPG (mmol/L) | -1.62 (0.106) | -2.08 (0.100) | -1.49 (0.105)
Statistical Analysis 1: Comparison: Dapaglifozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p = 0.374, Mixed Models Analysis; Mean Difference (Final Values) = -0.13, 95% CI 2-sided [-0.43 to 0.16]
Statistical Analysis 2: Comparison: Saxagliptin 5mg and Dapagliflozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.88 to -0.31]

5. Secondary Outcome: Time to Rescue
Description: The time to rescue (from first dose date after randomisation to start of rescue medication or discontinuation due to lack of glycaemic control) during the 52 week double blind treatment period
Time Frame: Over the 52 week treatment period
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
Weeks | NA [NA to NA] — Median time to rescue is not estimable due to the fact that less than 50% of patients had required rescue by the end of the treatment period (52 weeks). Cpnsequently the CI is not estimable either. | NA [NA to NA] — Median time to rescue is not estimable due to the fact that less than 50% of patients had required rescue by the end of the treatment period (52 weeks). Cpnsequently the CI is not estimable either. | NA [NA to NA] — Median time to rescue is not estimable due to the fact that less than 50% of patients had required rescue by the end of the treatment period (52 weeks). Cpnsequently the CI is not estimable either.
Statistical Analysis 1: Comparison: Dapaglifozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p = 0.777, Regression, Cox; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.67 to 1.35]
Statistical Analysis 2: Comparison: Saxagliptin 5mg and Dapagliflozin 10mg vs Glimepiride 1mg/2mg/4mg; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.36, 95% CI 2-sided [0.23 to 0.57]

6. Secondary Outcome: Number of Patients Rescued
Description: Number (%) of patients rescued.
Time Frame: Over the 52 week treatment period
Measure: Number; unit: Percentage of participants
Arm/Group | Dapaglifozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
Number analyzed (Participants) | 311 | 312 | 309
Percentage of participants | 18.6 | 8.3 | 21.4

ADVERSE EVENTS:
Time Frame: Adverse Events from signature of informed consent, enrolment, randomisation and throughout the 52 week treatment period and including the follow-up period. Serious Adverse Events from the time of informed consent.
Description: Safety Analysis Set (All randomised subjects who received at least 1 dose of study medication) N=313, 312, 312 for Dapa, Saxa+Dapa, Glim respectively. subjects excluded from the Safety Analysis Set (n=1,0, 1 for Dapa, Saxa+Dapa, Glim respectively) did not receive treatment.
Arm/Group | Dapagliflozin 10mg | Saxagliptin 5mg and Dapagliflozin 10mg | Glimepiride 1mg/2mg/4mg
All-Cause Mortality (participants affected / at risk) | 0/313 | 0/312 | 0/312
Serious Adverse Events (participants affected / at risk) | 39/313 | 22/312 | 35/312
Other Adverse Events (participants affected / at risk) | 29/313 | 31/312 | 37/312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg (N=313) | Saxagliptin 5mg and Dapagliflozin 10mg (N=312) | Glimepiride 1mg/2mg/4mg (N=312)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Bradyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 3 (3) | 2 (2)
Coronary artery occlusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Thyroid haemorrhage (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Vitritis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Micrococcus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Reiter's syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Brain stem infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Essential tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Vertebrobasilar insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Somatic symptom disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder prolapse (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral stenosis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Acquired phimosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dapagliflozin 10mg (N=313) | Saxagliptin 5mg and Dapagliflozin 10mg (N=312) | Glimepiride 1mg/2mg/4mg (N=312)
Nasopharyngitis (Infections and infestations) | 29 (40) | 31 (39) | 37 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-03-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT02471404/SAP_000.pdf
  • Study Protocol (2017-01-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT02471404/Prot_001.pdf